CLINICAL TRIAL: NCT00651092
Title: to Compare Two Well Popularized Methods of Inferior Nasal Turbinectomy
Brief Title: Inferior Submucosal Turbinectomy Versus Blunt Turbinectomy for Inferior Turbinate Hypertrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Dr nili segal, soroke university medical center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sor466208ctil
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Bilateral Inferior Turbinates Hypertrophy
Keywords: turbinectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Active Comparator): since the two methods of turbinectomy are in used on a regular basis there is no way to perform double blind study- both the surgeon and the patients are well aware of the operation they are about to go. we just compare several parameters in patients who are anyway about to undergo an operation in a specific method that is used by their surgeon
  Interventions: Procedure: bilateral nasal inferior turbinectomy
- A2 (Active Comparator): the resection of the inferior turbinates will be performed endonasally with an endoscopical instruments
  Interventions: Procedure: endoscopic submucosal resection of the inferior turbinates

INTERVENTIONS:
Procedure: bilateral nasal inferior turbinectomy — the operation is performed endonasally under general or local anesthesia, the inferior turbinates are resected and removed
  Other Names: inferior conchectomy
  Arms: A1
Procedure: endoscopic submucosal resection of the inferior turbinates — surgery of the inferior turbinates- endonasally with endoscopic instruments and by performing submucosal resection of the nasal turbinates
  Other Names: submucosal conchectomy
  Arms: A2

SUMMARY:
The aim of the study is to compare endoscopic submucosal inferior turbinectomy to blunt turbinectomy in terms of subjective and objective parameters.

DETAILED DESCRIPTION:
The two methods of nasal inferior turbinectomy are well popularized and in use for long periods of time. Endoscopic submucosal inferior turbinectomy is performed in our hospital and blunt turbinectomy is performed usually in privat clinics outside the hospital where there is no endoscopic equipment. We will examine both subjective (QOL questionaire) and objective parameters(rhinomanometry- a non invasive method to evaluate nasal airflow, saccharine test, nasal endoscopy) in our comparison of the outcome of these two methods.

ELIGIBILITY:
Inclusion Criteria:

* all patients above 18 years

Exclusion Criteria:

* can not answer a written questionaire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-05 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
quality of life | 1 year

SECONDARY OUTCOMES:
rhinomanometry, saccharine test, nasal endoscopy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: nili segal, md, Principal Investigator — soroka university medical center beer sheva israel

REFERENCES:
- [Result] Fradis M, Golz A, Danino J, Gershinski M, Goldsher M, Gaitini L, Malatskey S, Armush W. Inferior turbinectomy versus submucosal diathermy for inferior turbinate hypertrophy. Ann Otol Rhinol Laryngol. 2000 Nov;109(11):1040-5. doi: 10.1177/000348940010901109. PMID 11089995
- [Result] Williams HO, Fisher EW, Golding-Wood DG. 'Two-stage turbinectomy': sequestration of the inferior turbinate following submucosal diathermy. J Laryngol Otol. 1991 Jan;105(1):14-6. doi: 10.1017/s0022215100114707. PMID 1999659